CLINICAL TRIAL: NCT05996705
Title: Fatigue and Related Factors in Patients With Rheumatoid Arthritis
Brief Title: Fatigue in Patients With Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Gaziler Physical Medicine and Rehabilitation Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Yasin Demir, Associate professor, Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Other Study IDs: 40
Record Dates: First submitted 2023-08-10; First posted 2023-08-18 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Rheumatoid Arthritis
Keywords: fatigue; disease activity; rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Fatigue

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Determining the relationship of fatigue with some parameters — Determining the relationship of fatigue with physical function, pain values at rest and in motion, gender, age, pain, disease activity, gender and disease duration in RA patients.

SUMMARY:
Rheumatoid arthritis (RA) is a disease characterized by autoimmune systemic inflammatory polyarthritis, particularly affecting the joints of the hands. In addition to joint findings, extra-articular symptoms such as muscle pain, fatigue, fever and malaise are also common.

Fatigue is characterized by a feeling of extreme tiredness and persistent exhaustion. The prevalence of fatigue is between 14% and 15% in healthy adults. Although fatigue is common in patients with RA, it may remain in the background in clinical evaluation. The etiology of fatigue in RA is related to inflammation, pain, psychosocial factors and sleep disturbance, it has not been fully explained.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a disease characterized by autoimmune systemic inflammatory polyarthritis, particularly affecting the joints of the hands. In addition to joint findings, extra-articular symptoms such as muscle pain, fatigue, fever and malaise are also common.

Fatigue is characterized by a feeling of extreme tiredness and persistent exhaustion. The prevalence of fatigue is between 14% and 15% in healthy adults. Although fatigue is common in patients with RA, it may remain in the background in clinical evaluation. The etiology of fatigue in RA is related to inflammation, pain, psychosocial factors and sleep disturbance, it has not been fully explained.

There are various studies in the literature examining fatigue and factors associated with fatigue in patients with RA. This study aimed to contribute to the literature by determining the relationship of fatigue with physical function, pain values at rest and in motion, gender, age, pain, disease activity, gender and disease duration in RA patients.

ELIGIBILITY:
Inclusion Criteria:

* Age between 16-85 years
* Patients diagnosed with RA according to 2002 ACR-EULAR RA criteria.

Exclusion Criteria:

* Malignancy
* Neurological disease
* Major psychiatric disorder
* Thyroid disease
* Anemia and hypovitaminosis

Ages: 16 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients (38 males, 103 females) over 16 years of age who were diagnosed with RA according to the 2002 ACR-EULAR RA criteria.
Sampling Method: Non-Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2014-06-01 (Actual); Primary Completion 2016-03-01 (Actual); Study Completion 2016-03-01 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | through study completion, an average of one month
  Pain levels were evaluated with Visual Analogue Scale (VAS) (0 = no pain and 10 = the worst pain you can imagine) in motion and at rest.
Disease Activity Score-28 (DAS28) | through study completion, an average of one month
  Disease activity was assessed with the Disease Activity Score-28 (DAS28). Since the signs and symptoms of rheumatoid arthritis are very diverse, the DAS 28 scale, which evaluates disease activity in a combination of many parameters and has validity, was developed. DAS28 score below 3.2 is considered as low disease activity, between 3.2 and 5.1 as moderate disease activity, and above 5.1 as high disease activity. According to ACR criteria, a score below 2.6 is considered remission.
Health Assessment Questionnaire (HAQ) | through study completion, an average of one month
  Physical functioning and health-related quality of life were assessed with the Health Assessment Questionnaire (HAQ). The HAQ is approved by the American College of Rheumatology (ACR) for the assessment of physical function in rheumatoid arthritis. HAQ questions are given a score of 0 if the respondent can do them without any difficulty, 1 if they have some difficulty, 2 if they have a lot of difficulty and 3 if they cannot do them at all. The highest (worst) score in each domain is considered as the score of that domain. The HAQ score is obtained by summing the scores of the domains and dividing the total score by eight. If the HAQ score is 0-1, it is considered as mild-moderate disability, 1-2: moderate-severe disability, 2-3: severe-very severe disability.
Fatigue Symptom Inventory (FSI). | through study completion, an average of one month
  Fatigue was assessed with the Fatigue Symptom Inventory (FSI). It is a scale consisting of 14 questions in total. The FSI assesses maximum, minimum, average and current levels of fatigue over the past week on an 11-point scale (0: not tired at all, 10: extremely tired).

CONTACTS AND LOCATIONS:
Overall Officials: Gizem Kılınç Kamacı, MD, Principal Investigator — Specialist
Locations (1):
- Ankara Physical Medicine and Rehabilitation Training and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sandikci SC, Ozbalkan Z. Fatigue in rheumatic diseases. Eur J Rheumatol. 2015 Sep;2(3):109-113. doi: 10.5152/eurjrheum.2015.0029. Epub 2015 Sep 1. PMID 27708942
- [Background] Pollard LC, Choy EH, Gonzalez J, Khoshaba B, Scott DL. Fatigue in rheumatoid arthritis reflects pain, not disease activity. Rheumatology (Oxford). 2006 Jul;45(7):885-9. doi: 10.1093/rheumatology/kel021. Epub 2006 Jan 31. PMID 16449363